CLINICAL TRIAL: NCT02938507
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Immediate and Modified Release Formulations of Orally Administered Solabegron in Healthy Male Subjects
Brief Title: Evaluate the Safety, Tolerability and PK of Different Formulations of Orally Administered Solabegron in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Velicept Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: VEL-1001
Record Dates: First submitted 2016-10-12; First posted 2016-10-19 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Healthy Subjects, Overactive Bladder
Keywords: Overactive bladder, Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation 1 solabegron (Experimental): Subjects will receive formulation 1 solabegron doses in a single-blind, randomized, cross-over fashion in Periods 1 to 3.
  Interventions: Drug: Formulation 1 solabegron
- Formulation 2 solabegron (Experimental): Subjects will receive formulation 2 in a single-blind, randomized, cross-over fashion in Periods 1 to 3.
  Interventions: Drug: Formulation 2 solabegron

INTERVENTIONS:
Drug: Formulation 1 solabegron
  Arms: Formulation 1 solabegron
Drug: Formulation 2 solabegron
  Arms: Formulation 2 solabegron

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of different formulations of orally administered solabegron in healthy male subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of different formulations of orally administered solabegron in healthy male subjects. Eligible male subjects will be enrolled into 2 cohorts of 12 subjects each conducted in parallel. The study is a single blind (subjects), randomized, cross-over design in 3 study periods.

ELIGIBILITY:
Inclusion Criteria:

* Body weight greater than or equal to 50 kg, inclusive, and body mass index (BMI) 18.0 - 32.0 kg/m2, inclusive
* In good general health as determined by a thorough medical history and physical examination, ECG, vital signs, and clinical laboratory evaluation. Results of clinical laboratory tests must be without clinically significant abnormalities, including hematology, clinical chemistry and urinalysis.
* Adequate venous access to allow for repeated blood sampling
* Ability to understand and comply with the study requirements
* Provide written informed consent prior to any study procedure being performed (all subjects should be able to understand the informed consent form and any other documents that subjects are required to read).

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening physical examination, clinical laboratory tests, 12-lead ECG, or any other medical condition or circumstance which would make the subject unsuitable for participation in the study based on the Investigator's assessment
* Resting heart rate greater than or equal to 100 beats per minute (BPM) after 5 minutes rest (as above) at the screening visit
* QTcF interval (Fredericia's correction factor) greater than 450 msec (males subjects) at screening
* History of drug or other allergy, which, in the opinion of the Investigator, contraindicates their participation
* History of smoking, including e-cigarettes, within 3 months of the study and/or a positive urine cotinine at screening
* Regular alcohol consumption averaging ≥ 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of the first dose of study medication.
* Positive urine drug or alcohol test at screening
* Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for the study (e.g., due to expected study medication non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Eliot Ohlstein, PhD, Study Director — Velicept Therapeutics, Inc.

IPD SHARING:
Plan to Share IPD: No